CLINICAL TRIAL: NCT00986063
Title: A Multi-center, Double-blinded Randomized Trial for Genotype Based Personalized Prescription of Nevirapine
Brief Title: Genotype Based Personalized Prescription of Nevirapine
Acronym: GENPART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Surakameth Mahasirimongkol (Other)
Collaborators: Mahidol University (Other); Chulalongkorn University (Other); Thammasat University (Other); Srinakharinwirot University (Other); National Institutes of Health (NIH) (NIH); RIKEN (Other)
Responsible Party: Sponsor-Investigator, Surakameth Mahasirimongkol, Dr., Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GENPART
Record Dates: First submitted 2009-09-27; First posted 2009-09-29 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Nevirapine Induced Rash; Nevirapine Induced Hepatitis; HIV; Adverse Side Effects; AIDS; HIV Infections
Keywords: Nevirapine induced rash; Hepatitis; Pharmacogenomics; AIDS; HIV; treatment naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Hepatitis | interventions — Genetic Testing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator): AIDS patients taking care with standard of care
  Interventions: Other: 3TC/D4T/NVP or 3TC/AZT/NVP
- Genetic test (Experimental): AIDS patients who required highly active antiretroviral therapy(HAART) whom genotype status will be determined before initiation of HAART
  Interventions: Genetic: Genetic test for NVP induced rash

INTERVENTIONS:
Genetic: Genetic test for NVP induced rash — The genotype statuses that capable of predict the cutaneous side effects from nevirapine
  Arms: Genetic test
Other: 3TC/D4T/NVP or 3TC/AZT/NVP — Standard HAART for AIDS patients in Thailand
  Arms: Standard of care

SUMMARY:
Genetic tests has been suggested to reduce side effects related to Nevirapine(NVP), a commonly prescribed component of highly active antiretroviral therapy(HAART) in developing countries. This clinical trials is designed to determine the efficacy and the cost-effectiveness of this approach in the developing countries setting.

NVP-based HAART and efavirenz(EFV)-based HAART will be provided through Thai national universal health coverage. Information of the prescribed drug will be collected, and monitoring for the compliance with the prescribed highly active antiretroviral therapy will be conducted.

Outcome measurements:

The primary objective of this study is to evaluate the reduction in incidences of NVP associated cutaneous side effects by genotype based personalized prescription. The volunteers will be monitored for any solicited and non-solicited adverse effects for 6 months after drug administration, with first 6 weeks intensive monitoring for cutaneous adverse reactions. Laboratory safety profiles (Complete Blood Count(CBC), Alanine transaminase(ALT), Aspartate transaminase(AST), Blood Urea Nitrogen(BUN), creatinine, direct bilirubin, total bilirubin, lactate dehydrogenase, alkaline phosphatase) will be assessed during the intensive monitoring period (6 weeks).

Statistical Methods:

Descriptive statistics will be used to evaluate the conduct of the study. Analysis variables will include overall follow-up rate, drug compliance, and events of protocol violation.

Laboratory and safety data will be presented using comparative statistics for each study group and compared within and between groups using standard parametric or non-parametric comparison tests, i.e., McNemar's test or paired t-test as appropriate.

Comparison of rate of cutaneous adverse reaction, hepatitis and severe cutaneous adverse reaction(SCAR) will be made with chi-square test. Variable that shown significant different between the "standard of care" or control group and the "genetic test" or intervention group will adjusted for the final analysis with Poisson logistic regression.

The overall rate of adverse events in all participants will be monitored whether the rate of adverse events is lower than the predefined criteria. The extension of trial may be considered based on the rate of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (non-lactating and non-pregnant), aged between 18-70 years
* Written informed consent given after reading the volunteer information leaflet. Participation will be voluntary and volunteers will be fully informed of possible side effects. They will be advised that they are free to withdraw at any time.
* Has confirmed human immunodeficiency virus type 1 infection.
* Require antiretroviral based on standard practice guideline in Thailand.
* Adequate venous access
* Naïve to antiretroviral therapy standard clinical guideline in Thailand.
* Give consent to determine the genotype status

Exclusion Criteria:

* Women who are breast-feeding
* Participation in a study of any investigational drug where the study drug was received within the last 30 days
* Patients who received post or pre-exposure prophylaxis or single dose peripartum prevention incorporated of NVP will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To compare the incidences of nevirapine associated rashes in patients who are initiated nevirapine guided by genetic tests (genetic test group) and patients who are initiated nevirapine using standard of care approach (control group). | 6 months

SECONDARY OUTCOMES:
To determine the cost-effectiveness of genotyped based personalized prescription of nevirapine. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Somnuek Sungkanuparph, MD, Principal Investigator — Infectious disease Unit, Department of Internal Mediciine, Faculty of Ramathibodi Medical School, Mahidol University
Locations (1):
- Division of Infectious Diseases, Department of Medicine, Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok, Thailand